CLINICAL TRIAL: NCT01449656
Title: A Randomized Trial Comparing the Laryngeal Mask Airway-SupremeTM With the Laryngeal Mask Airway-ProsealTM in Children
Brief Title: A Comparison of the Laryngeal Mask Airway (LMA) Proseal and LMA Supreme in Children
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Principal investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: PLMA vs SLMA
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Children
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LMA proseal
  Interventions: Device: LMA Proseal: control device
- LMA Supreme
  Interventions: Device: LMA Supreme: comparison device

INTERVENTIONS:
Device: LMA Proseal: control device — LMA Proseal will be placed in children weighing 10-20kg based on a computer generated randomization
  Other Names: laryngeal mask airway
  Groups: LMA proseal
Device: LMA Supreme: comparison device — LMA Supreme will be placed in children weighing 10-20kg based on a computer generated randomization
  Other Names: laryngeal mask airway
  Groups: LMA Supreme

SUMMARY:
The aim of this randomized prospective study is to compare two laryngeal mask airways with a provision for evacuation of gastric contents, the LMA Proseal and The investigators hypothesize that airway leak pressures with the LMA Proseal will be significantly different (higher) when compared with the LMA Supreme.

DETAILED DESCRIPTION:
The goal of this study is to compare the LMA Proseal and LMA Supreme in children having surgery. The investigators hypothesize that the airway leak pressures with the LMA Proseal will be superior to the LMA Supreme. Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached. The ease of placement of the device and gastric tube, fiberoptic grade of laryngeal view, feasibility of use during positive pressure ventilation, and complications (airway related, gastric insufflation, trauma) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia using a supraglottic airway device
* weight 10-20 kg
* age 6 months-6 years

Exclusion Criteria:

* ASA class IV, V Emergency procedures
* History of a difficult airway
* Active gastrointestinal reflux
* Active upper respiratory tract infection

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children weighing 10 to 20 kg undergoing surgical or medical procedures under anesthesia requiring a supraglottic airway device
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Airway Leak Pressure | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached when fresh gas flow is delivered at 3L/min when the pressure limiting valve is closed completely.

SECONDARY OUTCOMES:
Time to secure the airway | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  From picking up the airway device to bilateral chest expansion and presence of ETCO2
Number of attempts to place the device | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  number of attempts needed for successful placement will be recorded (maximum of 3 attempts will be considered as a failure)
Fiberoptic grade of laryngeal view | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The laryngeal alignment through the devices will be graded using an established scoring system
Gastric insufflation | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The presence of gastric insufflations will be assessed during leak pressure testing by using epigastric auscultation
Ease of gastric tube placement | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The ease of gastric placement will be timed and assessed using a subjective scale
Fiberoptic view through the gastric tube | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The view through the gastric drain tube of the LMA supreme will be assessed and graded using an established scoring system
feasibility of positive pressure ventilation | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Peak inspiratory pressure and tidal volumes will be recorded. Maximum peak inspiratory pressure will be the airway leak pressure was determined for each patient
Quality of the airway | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The quality of hands free anesthesia will be assessed during maintenance of anesthesia using a previously described scale
Adverse effects | Participants will be followed for the duration of anesthesia and 24 hours postoperatively
  complications such as oxygen desaturations, mucosal trauma, reflex activation of the airway, sore throat, dysphonia will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Childrens Memorial Hospital
Locations (1):
- Childrens Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Trevisanuto D, Parotto M, Doglioni N, Ori C, Zanardo V, Micaglio M. The Supreme Laryngeal Mask Airway (LMA): a new neonatal supraglottic device: comparison with Classic and ProSeal LMA in a manikin. Resuscitation. 2012 Jan;83(1):97-100. doi: 10.1016/j.resuscitation.2011.07.032. Epub 2011 Aug 11. PMID 21839703
- [Background] Seet E, Rajeev S, Firoz T, Yousaf F, Wong J, Wong DT, Chung F. Safety and efficacy of laryngeal mask airway Supreme versus laryngeal mask airway ProSeal: a randomized controlled trial. Eur J Anaesthesiol. 2010 Jul;27(7):602-7. doi: 10.1097/eja.0b013e32833679e3. PMID 20540172
- [Background] White MC, Cook TM, Stoddart PA. A critique of elective pediatric supraglottic airway devices. Paediatr Anaesth. 2009 Jul;19 Suppl 1:55-65. doi: 10.1111/j.1460-9592.2009.02997.x. PMID 19572845